CLINICAL TRIAL: NCT06551038
Title: Evaluating Primary Suicide Prevention in Adolescents With Risk Factors
Acronym: ESPAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephanie Baggio (Other)
Responsible Party: Sponsor-Investigator, Stephanie Baggio, Associate Professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-01208
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Suicide Prevention
Keywords: Suicide; Primary prevention; Vulnerable adolescents; Psychological distress
MeSH Terms: conditions — Suicide Prevention; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary suicide prevention intervention (Experimental): The framework of the primary suicide prevention intervention is psychoeducation. The intervention lasts for 90 minutes and is conducted in groups of 5 to 15 (on average 10) participants. It provides general information on suicidal behaviors, information about facts and myths about suicide, identification of risk factors and warning signs of suicidal behaviors, and information on ways to seek for help and get support for themselves and others in the canton. The intervention includes a lecture, group discussions based on case examples, and a quiz on facts and myths about suicide. It is conducted by a trained staff member with the support of a psychologist trained in suicide prevention for children and adolescents. It follows a standardized format.
  Interventions: Behavioral: Primary suicide prevention intervention
- Art-based control intervention (Active Comparator): The control intervention will be an art-based activity, a workshop on slam poetry. At the end of the study, participants will get a flyer containing information on suicide prevention with the participants of the control group. Therefore, they will have a low-threshold intervention.
  Interventions: Behavioral: Art-based control intervention

INTERVENTIONS:
Behavioral: Primary suicide prevention intervention — Psychoeducation workshop
  Arms: Primary suicide prevention intervention
Behavioral: Art-based control intervention — Slam poetry workshop
  Arms: Art-based control intervention

SUMMARY:
Suicide is one of the main causes of death among teenagers. Because it is preventable, primary prevention of suicide has become a public health priority, with encouraging results in promoting suicide awareness and reducing suicidal thoughts among adolescents. However, the lack of studies conducted among vulnerable populations (i.e., marginalised, disengaged and disadvantaged) is a major gap, even though these populations present an increased risk of suicidal behaviour.

The aim of this project is to test the effectiveness of a brief primary suicide prevention intervention for vulnerable adolescents, using a randomised controlled trial. Vulnerable adolescents include those 1) detained in juvenile detention centres, 2) at risk of dropping out of school, 3) undergoing treatment for psychiatric disorders, 4) belonging to a sexual or gender diversity, 5) affected by chronic conditions, or 6) with relational/familial problems. The main aim is to test the effectiveness of the intervention on a composite measure of suicide awareness, psychological distress and suicidal thoughts. The project will also explore other issues that present challenges for vulnerable populations: access to primary suicide prevention and non-response bias. The study will provide relevant results to address the current lack of high-quality evidence for primary suicide prevention in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Vulnerable adolescents defined as being: 1) detained in juvenile detention centers, 2) disconnected from school, 3) in treatment for psychiatric disorders, 4) belonging to a sexual or gender minority, 5) affected by chronic conditions, or 6) with relational/familial problems.
* Age 14 to 25 years old.
* Good knowledge of French.
* Accepting to sign the informed consent.

Exclusion Criteria:

* The medical/educational staff considers that the intervention will interfere with appropriate management of acute psychiatric disorder or may cause harm to self or other.
* Being enrolled in another suicide prevention intervention during the study period.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite measure of suicide awareness | One-week post-baseline
  Nine-item perceived suicide awareness scale (PSAS-9), assessed on a 5-point scale, score ranging from 0 to 36, with a higher score indicating a higher suicide awareness

SECONDARY OUTCOMES:
Composite measure of suicide awareness | Three-month post-baseline
  Nine-item perceived suicide awareness scale (PSAS-9), assessed on a 5-point scale, score ranging from 0 to 36, with a higher score indicating a higher suicide awareness
Knowledge on suicide | One-week post-baseline; three-month post-baseline
  Literacy of Suicide Scale (LOSS), 12 binary (true/false) questions, score ranging from 0 to 12, with a higher score indicating higher knowledge on suicide
Knowledge of local resources | One-week post-baseline; three-month post-baseline
  Self-developed scale on local resources, 6 binary (true/false) questions, score ranging from 0 to 6, with a higher score indicating higher knowledge of local resources
Suicidal thoughts | One-week post-baseline; three-month post-baseline
  Suicidal Ideation Attributes Scale (SIDAS), 10 questions assessed on a 5-point scale, with a score ranging from 0 to 50. A higher score indicates a higher level of suicidal thoughts.
Psychological distress | One-week post-baseline; three-month post-baseline
  Kessler Psychological Distress scale (K-6), 6-item scale is assessed on a 5-point scale, with a score ranging from 0 to 24. A higher score indicates a higher level of psychological distress.
Access to primary suicide prevention | Baseline
  Self-developed scale on primary suicide prevention training, 3 questions combined in a binary indicator (yes/no)
Attrition | Three-month post-baseline
  Percentage of participants who drop out, continuous variable (0-100), with a higher percentage indicating a higher level of attrition

OTHER OUTCOMES:
Number of participants with serious adverse events (safety outcome) | One-month post baseline
  Death, life-threatening event, and hospitalisation
Number of participants with adverse events (safety outcome) | One-month post baseline
  Scarification, insomnia, appetite problems, substance use, and para-suicidal endangerment behaviors identified and reported by the local team
Self-reported distress (safety outcome) | One-week post-baseline
  Composite outcome with two questions from Bailey et al. (2017, https://https://doi.org/10.1027/0227-5910/a000465) related to the distressing and pleasurable nature of the intervention, assessed on a 5-point scale, score ranging from 0 to 8, a higher score indicating higher self-reported distress

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Baggio, Prof., Principal Investigator — Institute of Primary Health Care (BIHAM), University of Bern
Locations (19):
- Switzerland (19):
  - Dialogai et Totem, Geneva, Canton of Geneva
  - Programme ForMe (anciennement SEMO) et dispositif ProPULSE, Plan-les-Ouates, Canton of Geneva
  - Centre de Détention et d'Observation La Clairière, Vernier, Canton of Geneva
  - Programme Intégration et Formation Professionnelle, Vernier, Canton of Geneva
  - Agnodice, Lausanne, Canton of Vaud
  - Vogay, Lausanne, Canton of Vaud
  - Centre Thérapeutique de Jour pour Adolescents, Lausanne, Canton of Vaud
  - Unité de Soins Psychiatriques Fermée pour Mineurs, Lausanne, Canton of Vaud
  - Établissement de Détention pour mineurs et jeunes adultes Les Léchaires, Palézieux, Canton of Vaud
  - Centre éducatif fermé de Pramont, Sierre, Valais
  - CAP Formations, Cité des Métiers, Geneva
  - Unité de Liaison Ambulatoire et Hospitalière, Service de psychiatrie de l'enfant et de l'adolescent, HUG, Geneva
  - Foyers de Gilly, Grand-Lancy
  - Foyer de Chailly, Lausanne
  - Ren'Fort, Lausanne
  - Foyer La Pommeraie, Lonay
  - Service des Parcours Individualisé, Onex
  - Le Repuis, Petit Lancy
  - Astural, Parcours A2mains, Thônex

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on https://www.swissubase.ch.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the main results of the study
Access Criteria: Upon approval from the principal investigator

REFERENCES:
- [Derived] Baggio S, Bailey E, Edan A, Heller P, Kapp C, Lambert N, Michaud L, Mundt AP, Nsingi N, Perez S, Peregalli S, Piguet C, Piotrowski C, Prutyanova Y, Rumley M, Sapin M, Urben S, Iglesias K. Evaluating primary suicide prevention in adolescents with risk factors (ESPAIR): study protocol for a cluster-randomized controlled trial. Trials. 2025 Nov 24;26(1):537. doi: 10.1186/s13063-025-09266-y. PMID 41286939